CLINICAL TRIAL: NCT01587911
Title: Characterization of the Physiological and Subjective Satiety Response to Preloads Varying in Bioactive Dairy Proteins
Brief Title: Casinomacropeptide and Satiety
Acronym: CMP2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: 200614016
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Lack of Satiety; Excess Intake of Macronutrients; Appetite Disorders
Keywords: Satiety; Food intake regulation; Appetite regulation; Dairy Protein
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Whey; Cytidine Monophosphate; cyclopropapyrroloindole; Caseins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Whey protein (Active Comparator): Complete whey protein.
  Interventions: Other: Whey
- Whey-CMP (Active Comparator): Complete whey protein missing the CMP (aka GMP) portion of the peptide.
  Interventions: Other: Whey-CMP
- Control (Placebo Comparator): Placebo preload control, matched for energy.
  Interventions: Other: Control
- CMP (casinomacropeptide) (Active Comparator): Small peptide cleaved from complete whey protein.
  Interventions: Other: CMP
- MPI (Active Comparator): Complete milk protein.
  Interventions: Other: MPI
- CPI (casein) (Active Comparator): Preload containing casein.
  Interventions: Other: CPI

INTERVENTIONS:
Other: Whey — Preload containing complete whey protein.
  Other Names: Whey.
  Arms: Whey protein
Other: Whey-CMP — Preload containing complete whey protein which is missing the CMP/GMP portion of the protein.
  Arms: Whey-CMP
Other: Control — Preload control matched for energy to the other 5 preloads.
  Arms: Control
Other: CMP — Preload containing the CMP (casinomacropeptide) portion cleaved from complete whey protein.
  Other Names: casinomacropeptide
  Arms: CMP (casinomacropeptide)
Other: MPI — Preload containing whole milk protein.
  Other Names: Whole milk protein
  Arms: MPI
Other: CPI — Preload containing sodium caseinate.
  Other Names: Casein
  Arms: CPI (casein)

SUMMARY:
Assessing 5 different milk derived proteins versus placebo for appetite regulation and satiety, delivered via shake vehicle.

DETAILED DESCRIPTION:
Assessing 5 different milk derived proteins versus placebo for appetite regulation and satiety, delivered via shake vehicle. Subjects will attend a 5 hour post-prandial study day. Subjects will keep food records 1 and 3 days prior to study visit, day of visit, and day after visit; food to be weighed using study provided dietary scale.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Unrestrained (score ≤ 10 on the Eating Inventory (EI) questionnaire, Stunkard and Messick 1985)
* Women
* 18 years of age
* Consume a low/moderate protein diet (12-20% protein energy).
* Meet BMI criteria of 19 to 24 kg/m2 OR 29 to 34 kg/m2, inclusive.

Exclusion Criteria:

* Women who score ≥ 10 on the Beck Depression Inventory (BDI, Beck and Beamesdorfer 1974)
* Women who score ≥ 30 on Eating Attitudes Test (EAT, Garner and Garfinkel 1979),
* Have current or past (previous 1 year) medical conditions that may interfere with any of the outcomes of this study.
* Weigh less than 110 lbs
* Are currently or have been modifying diet or exercise patterns to gain or lose weight in previous 60 days
* Have unstable body weight (fluctuations of ≥ 5 kg in 60 day period)
* Are excessive exercisers or trained athletes
* Taking any medications that would affect appetite or any other study-described endpoint will also be excluded.
* Allergies or intolerances to foods consumed in the study.
* Smoker
* Pregnant/lactation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-05; Primary Completion 2009-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Post-prandial satiety | 6 hours
  Blood biochemical markers of appetite regulation.
Post-prandial satiety | 6 hours
  Assessing biobehavioral aspects of appetite regulation through VAS.

SECONDARY OUTCOMES:
Extended satiety | 48 hours
  Utilizing self reported food intake, looking for changes associated with the different proetin compositions of the shakes.

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, PhD, MS, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis (Ragle Human Nutrition Research Center), Davis, California, United States